CLINICAL TRIAL: NCT07348250
Title: An Open-label Study to Evaluate Brain α-Synuclein Deposition Using Positron Emission Tomography (PET) and [18F]MK-0947 in Patients With Parkinson's Disease
Brief Title: Open-label Study to Evaluate Brain α-Synuclein Deposition Using PET and [18F]MK-0947 in Parkinson's Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Invicro (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: MK-0947 PN001
Record Dates: First submitted 2025-12-29; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease (PD); Parkinson's Disease; Parkinson's Disease (Disorder)
Keywords: alpha-synuclein; α-synuclein; Neurodegeneration; MK-0947
MeSH Terms: conditions — Parkinson Disease; Parkinson Disease 4, Autosomal Dominant Lewy Body; Nerve Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 - Brain Imaging (Experimental): Participants receive [18F]MK-0947 for PET imaging of the brain.
  Interventions: Drug: [18F]MK-0947
- Part 2 - Dosimetry (Experimental): Healthy participants receive [18F]MK-0947 for whole-body dosimetry.
  Interventions: Drug: [18F]MK-0947

INTERVENTIONS:
Drug: [18F]MK-0947 — PET radiopharmaceutical selective for α-synuclein, administered IV at doses up to 10 mCi.
  Other Names: MK-0947

SUMMARY:
This clinical study is being conducted to learn more about a new imaging drug called [18F]MK-0947, which is designed to help doctors see changes in the brain related to Parkinson's disease (PD). PD is a condition that affects movement, balance, and thinking. The drug works with a type of scan called PET (Positron Emission Tomography) to show areas of the brain where a protein called α-synuclein builds up. This buildup is linked to PD and other brain disorders.

The main goal of this study is to find out if [18F]MK-0947 is safe for people and if it works well to show α-synuclein in the brain. The study will also look at how the drug moves through the body and how much radiation it gives off. Researchers hope this information will help develop better tools for diagnosing PD and tracking how it changes over time.

Who can join? Adults who have PD or who are healthy may be able to take part. Participants will have screening tests to make sure they qualify.

What does participation involve? People in the study will have PET scans, blood tests, and other safety checks. Some participants will also have an MRI scan. The study is divided into two parts: Part 1 looks at how the drug works in the brain of PD patients and healthy elderly participants, and Part 2 measures radiation levels in healthy participants.

Why is this important? There is currently no cure for PD, and better imaging tools could help researchers develop new treatments. By joining this study, participants will help advance research that may improve care for people with PD and similar conditions in the future.

DETAILED DESCRIPTION:
This Phase 1, open-label study will evaluate the safety, pharmacokinetics, and imaging characteristics of [18F]MK-0947, a novel PET tracer targeting α-synuclein pathology in Parkinson's disease (PD). The study consists of two parts: Part 1 includes PD and healthy elderly participants for brain imaging using standard and high-resolution PET scanners; Part 2 includes healthy participants for whole-body dosimetry to estimate radiation exposure. Imaging sessions will involve dynamic PET scans lasting up to 2 hours, arterial or venous blood sampling for kinetic modeling, and MRI for anatomical co-registration. Safety assessments include vital signs, ECGs, laboratory tests, and adverse event monitoring. The investigational tracer will be administered intravenously at doses up to 10 mCi, with strict adherence to radiation safety guidelines. Data will be analyzed using compartmental and graphical modeling approaches to derive quantitative metrics such as SUV, SUVR, VT, and DVR. This study aims to establish proof of concept for [18F]MK-0947 as a biomarker for α-synuclein pathology, supporting future therapeutic trials and advancing diagnostic capabilities for synucleinopathies.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study procedures
* Women of childbearing potential: abstinent or use 2 contraception methods (one barrier) during study and 90 days post last injection
* Men: use 2 contraception methods and refrain from sperm donation during study and 90 days post last injection
* PD & HE participants: Age 40-80 years; HP participants: Age 18-50 years
* Adequate circulation and normal clotting for arterial cannulation (if applicable)
* HE participants: no neurological disorder, no first-degree relative with idiopathic PD
* HP participants: healthy with no clinically relevant findings

Exclusion Criteria:

* Unwilling or unable to provide informed consent
* Clinically significant hepatic, renal, cardiovascular, pulmonary, or systemic illness
* Pregnant or breastfeeding
* Contraindication to PET or MRI procedures (e.g., implants, claustrophobia)
* History of severe allergic reactions to PET tracers or related compounds
* Current or prior participation in investigational drug study within 30 days
* Any condition that may interfere with study conduct or participant safety

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety of [18F]MK-0947: Incidence of Adverse Events | Up to 4 months
  Incidence of adverse events (AEs) following administration
Safety of [18F]MK-0947: Radiation absorbed dose estimates | 4 months
  Radiation absorbed dose estimates following administration derived from PET imaging and dosimetry calculations.

SECONDARY OUTCOMES:
Brain uptake of [18F]MK-0947 | Up to 36 days
  Quantitative assessment of [18F]MK-0947 uptake in brain regions measured by PET imaging.
Model-derived Pharmacokinetics of [18F]MK-0947 | Up to 36 days
  Pharmacokinetic parameters of [18F]MK-0947 derived from dynamic PET imaging and plasma input functions.

CONTACTS AND LOCATIONS:
Locations (1):
- Invicro (dba Perceptive), New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided